CLINICAL TRIAL: NCT00419211
Title: "Fit Pregnancy": A Transtheoretical-Model Based Intervention Designed To Increase Physical Activity and Maternal Well-Being During Pregnancy
Brief Title: An Intervention Study to Increase Physical Activity and Maternal Well-being During Pregnancy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Deborah Da Costa, Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A06-B25-06A
Record Dates: First submitted 2007-01-04; First posted 2007-01-08 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Pregnancy; Depression
Keywords: Pregnancy, Exercise, Depression
MeSH Terms: conditions — Depression; Motor Activity | interventions — Exercise

ARMS (2):
- Lifestyle counseling (Experimental): Tailored exercise program
  Interventions: Behavioral: Exercise
- No Intervention (No Intervention): Usual care group

INTERVENTIONS:
Behavioral: Exercise — Tailored exercise program
  Arms: Lifestyle counseling

SUMMARY:
To refine, implement and evaluate a motivationally-tailored exercise intervention for increasing physical activity and mental health during pregnancy and the postpartum.

DETAILED DESCRIPTION:
Pregnancy appears to pose a further barrier to exercise, as women remain inactive or cease to exercise all together. Yet, regular physical activity during pregnancy in healthy women has been shown to be safe and positively associated with physical and psychological health benefits. To date interventions to promote physical activity have not targeted pregnant women. We are proposing to pilot the first study to evaluate a theory-derived intervention designed to promote physical activity during pregnancy. We anticipate that pregnant women assigned to the motivationally-tailored exercise intervention will show a significant increase in physical activity from baseline at the post-treatment follow-up (32 weeks gestation). We expect that the motivationally-tailored intervention will positively influence physical and mental health status during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant

Exclusion Criteria:

* Regular participation in moderate intensity exercise for at least 30 minutes, 3 or more times a week at the time of study entry
* Contraindications for participating in exercise during pregnancy as outlined by the SOGC/CSEP clinical practice guidelines
* Inability to communicate in either English or French.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2007-01; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Physical Activity Level | post-intervention and 3 months after felivery
Depressed Mood | post-intervention and 3 months following delivery
Health related quality of life | post-intervention and 3 months following delivery

SECONDARY OUTCOMES:
state anxiety | post-intervention and 3 months following delivery
sleep quality | post-intervention and 3 months following delivery
fatigue levels | post-intervention and 3 months following delivery
exercise stage of change | post-intervention and 3 months following delivery
self-efficacy for exercise | post-intervention and 3 months following delivery
social support for exercise | post-intervention and 3 months following delivery

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Da Costa, PhD, Principal Investigator — McGill University
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada